CLINICAL TRIAL: NCT00253591
Title: Randomised Phase II/III Trial of Induction Chemotherapy Followed by Continuous Hyperfractionated Accelerated Radiotherapy (CHART) Versus CHART Alone in Patients With Inoperable Non-Small Cell Lung Cancer
Brief Title: Radiation Therapy With or Without Vinorelbine and Cisplatin in Treating Patients With Stage I, Stage II, or Stage III Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000449972; MRC-LU23; EU-20535; EU-INCH-20535; EudraCT-2004-004438-15
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-07

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Vinorelbine; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: vinorelbine tartrate
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as vinorelbine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether giving radiation therapy together with vinorelbine and cisplatin is more effective than radiation therapy alone in treating non-small cell lung cancer.

PURPOSE: This randomized phase II/III trial is studying how well giving radiation therapy together with vinorelbine and cisplatin works and compares it to radiation therapy alone in treating patients with stage I, stage II, or stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall survival of patients with stage I-III non-small cell lung cancer treated with vinorelbine, cisplatin, and continuous hyperfractionated accelerated radiotherapy (CHART) vs CHART alone.

Secondary

* Compare the response, progression-free survival, and quality of life of patients treated with these regimens.
* Compare the toxic effect of these regimens in these patients.
* Compare the cost effectiveness of these regimens in these patients.
* Compare the local and distant control in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo continuous hyperfractionated accelerated radiotherapy (CHART) 3 times a day for 12 consecutive days.
* Arm II: Patients receive vinorelbine IV over 5-10 minutes on days 1 and 8 and cisplatin IV over 2 hours on day 1. Treatment repeats every 21 days for 3 courses in the absence of disease progression or unacceptable toxicity. Beginning 4-6 weeks later, patients undergo CHART as in arm I.

Quality of life is assessed periodically.

After completion of study treatment, patients are evaluated periodically for at least 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage I-III non-small cell lung cancer

  * Inoperable or patient refuses surgery
* Disease can be encompassed within the radical radiotherapy treatment volume

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-1

Life expectancy

* More than 3 months

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 1.5 times upper limit of normal

Renal

* Glomerular filtration rate > 60 mL/min

Cardiovascular

* No uncontrolled arterial hypertension
* No ischemic heart disease

Pulmonary

* FEV_1 > 50% of predicted OR
* DLCO > 50% of predicted

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior or current malignancy that would preclude study treatment
* Medically stable
* No unstable diabetes
* No infection
* No hypercalcemia

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
Progression-free survival
Toxicity
Response (complete or partial response)
Cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hatton, MD, Study Chair — Cancer Research Centre at Weston Park Hospital
Locations (20):
- United Kingdom (20):
  - Wansbeck General Hospital, Ashington, England
  - Bristol Haematology and Oncology Centre, Bristol, England
  - Cheltenham General Hospital, Cheltenham, England
  - Derbyshire Royal Infirmary, Derby, England
  - University Hospital of North Durham, Durham, England
  - Queen Elizabeth Hospital, Gateshead, England
  - Northern Centre for Cancer Treatment at Newcastle General Hospital, Newcastle upon Tyne, England
  - Mount Vernon Cancer Centre at Mount Vernon Hospital, Northwood, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Kings Mill Hospital, Nottinghamshire, England
  - Churchill Hospital, Oxford, England
  - Cancer Research Centre at Weston Park Hospital, Sheffield, England
  - Great Western Hospital, Swindon, England
  - Worcester Royal Hospital, Worcester, England
  - Yeovil District Hospital, Yeovil, England
  - Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Crosshouse Hospital, Kilmarnock, Scotland
  - Velindre Cancer Center at Velindre Hospital, Cardiff, Wales
  - Llandough Hospital, Llandough, Wales
  - Royal Gwent Hospital, Newport Gwent, Wales